CLINICAL TRIAL: NCT00774696
Title: The Objective of This Study is to Compare the Relative Bioavailability of Clarithromycin 500 mg Tablets (Ranbaxy Laboratories Limited) With That of BIAXIN® 500 mg Tablets in Healthy, Adult Subjects Under Non-Fasting Conditions.
Brief Title: Bioequivalence Study of Clarithromycin 500 mg Tablets Under Non-Fasting Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ranbaxy Laboratories Limited (Industry)
Responsible Party: Tausif Monif, Ranbaxy Research Laboratories
Organization: Ranbaxy Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: B025512
Record Dates: First submitted 2008-10-15; First posted 2008-10-17 (Estimated); Last update posted 2008-10-17 (Estimated); Status verified 2008-10

CONDITIONS: Healthy
Keywords: Bioequivalence study of clarithromycin
MeSH Terms: interventions — Clarithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Clarithromycin 500 mg Tablets
  Interventions: Drug: clarithromycin 500mg tablets
- 2 (Active Comparator): BIAXIN® 500 mg tablets
  Interventions: Drug: clarithromycin 500mg tablets

INTERVENTIONS:
Drug: clarithromycin 500mg tablets

SUMMARY:
The objective of this study is to compare the relative bioavailability of clarithromycin 500 mg tablets (Ranbaxy Laboratories Limited) with that of BIAXIN® 500 mg tablets in healthy, adult subjects under non-fasting conditions.

DETAILED DESCRIPTION:
The study was conducted as an open label, balanced, randomised, two-treatment, two-period, two-sequence, single-dose, crossover , bioavailability study on clarithromycin formulations comparing clarithromycin 500mg tablets of Ranbaxy Laboratories with Biaxin® tablets 500mg (containing clarithromycin 500 mg)in healthy, adult, human, male subjects under fed conditions Subjects were given a standardized meal starting 30 minutes before their assigned dosing time consisting of one buttered English muffin, one fried egg, one slice of American cheese, one slice of Canadian bacon, 2.45 ounces of hash brown potatoes, six fluid ounces of orange juice, and eight fluid ounces of whole milk.

A single oral dose of clarithromycin 500mg was administered during each period under supervision of a trained Medical Officer.

During the course of study, the safety parameters including vital signs, physical examination, medical history, clinical laboratory and safety tests (haematology, biochemical parameters) were assessed and, clinical laboratory safety tests (hematology & biochemical parameters) were performed again at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Source of Subjects: Non-institutionalized subjects consisting of members of the community at large.
2. Characterization of Study Group

   * All subjects selected for this study will be at least 18 years of age. Female subjects must be unable to become pregnant (postmenopausal for at least 1 year, or surgically sterile).
   * Each subject shall be given a general physical examination within 28 days of initiation of the study. Such examinati°n includes, but is not limited to, blood pressure, general observations, and history.

Each female subject will be given a serum pregnancy test as part of the pre-study screening process. At the end of the study, the subjects will have an exit evaluation consisting of interim history, global evaluation, and clinical laboratory measurements. Adequate blood and urine samples should be obtained within 28 days before beginning of the first period and at the end of the trial for clinical laboratory measurements.

Drags of Abuse Screen: pre-study and at check-in each study period subjects will be selected if all above are normal. Electrocardiograms of all participating subjects will be recorded before initiation of the study and filed with each Subject's case report forms.

Exclusion Criteria:

1. Subjects with a history of chronic alcohol consumption (during past 2 years), drug addiction, or serious gastrointestinal, renal, hepatic or cardiovascular disease, tuberculosis, epilepsy, asthma(during past 5 years), diabetes, psychosis or glaucoma will not be eligible for this study.
2. Subjects whose clinical laboratory test values are greater than 20% outside the normal range may be retested. If the clinical values are outside the range on retesting, the subject will not be eligible to participate in the study unless the clinical investigator deems the result to not be significant.
3. Subjects who have a history of allergic responses to theclass of drag being tested (including any penicillin product) should be excluded from the study.
4. All subjects will have urine samples assayed for the presence of drugs of abuse as part of the clinical laboratory screening procedures at check-in each study period. Subjects found to have urine concentrations of tested will not be allowed to participate.
5. Subjects should not have donated blood or plasma for at least (30) days prior to first dosing of the study.

g. Female subjects who are pregnant or who are able (women child bearing potential) to become pregnant during the study not be allowed to participate.

h. All female subjects will be screened for pregnancy at check in each study period. Subjects with positive pr inconclusive results will be withdrawn from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24
Dates: Start 2002-12; Primary Completion 2002-12 (Actual); Study Completion 2003-02 (Actual)

PRIMARY OUTCOMES:
Bioequivalence

CONTACTS AND LOCATIONS:
Locations (1):
- Gateway Medical Research Inc., Saint Charles, Missouri, United States

REFERENCES:
- See also: Related Info — http://clinicalstudies.ranbaxy.com
- See also: Related Info — http://www.fda.gov/opacom/7alerts.html
- See also: Related Info — http://dailymed.nlm.nih.gov/dailymed/about.cfm